CLINICAL TRIAL: NCT06305156
Title: Protocol-optimization in Computed Tomography for the Quantification of Bone Mineral Density (BMD)
Brief Title: Protocol Optimization in CT for the Quantification of BMD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hatem Alkadhi (Other)
Responsible Party: Sponsor-Investigator, Hatem Alkadhi, Senior Attending Physician, Vice Director of the Institute, Institute for Diagnostic and Interventional Radiology, University of Zurich
Organization: University of Zurich (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CT_BMD_1
Record Dates: First submitted 2024-02-22; First posted 2024-03-12 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Osteoporosis, Osteopenia; Bone Loss
MeSH Terms: conditions — Osteoporosis; Bone Diseases, Metabolic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Bone mineral density CT vs DXA (Other): Single arm study, all participants receive CT and DXA.
  Interventions: Diagnostic Test: Bone Mineral Density quantification

INTERVENTIONS:
Diagnostic Test: Bone Mineral Density quantification — In the first visit, participants receive clinically indicated CT scan, where bone mineral density will be derived.
  In a second, study related visit, participants will receive a DXA scan for bone mineral quantifications.

SUMMARY:
Bone mineral density is an important measurement to detect osteoporosis.

The goal of this clinical trial is to compare bone mineral density measurements in CT examinations and DXA scans. The main question it aims to answer is:

* How good is the measurement of bone mineral density in the new photon-counting CT in comparison to DXA
* How can we optimize the CT scan for bone mineral density

Participants will undergo:

* Clinically indicated CT scan on day of inclusion
* Study related DXA scan on a separate appointment

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent signed by the subject
* Referral to a regular clinically indicated CT examination covering the lumbar area (e.g., Abdomen, Thorax + Abdomen, Neck + Thorax +Abdomen)
* Informed written and oral consent (interpreter present in case of foreign language patients)
* No contraindication to the clinically indicated CT examination

Exclusion Criteria:

* Patients < 18 years
* Pregnant women
* Vulnerable subjects
* Contraindications to the clinically indicated CT scan
* Multiple Myeloma
* Diffuse bone metastasis
* Fixateur interne in the lumbar spine
* Kyphoplasty in the lumbar spine
* Enterally administrated contrast agent
* Obtaining informed consent is not possible
* Withdrawal of consent orally or in writing
* Inability to follow the procedures of the investigation, e.g., due to language problems, psychological disorders, dementia, etc. of the subject
* Immobility (patients confined to a wheelchair or to bed)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 167 (Actual)
Dates: Start 2024-03-13 (Actual); Primary Completion 2025-12-19 (Actual); Study Completion 2025-12-19 (Actual)

PRIMARY OUTCOMES:
Bone mineral density CT | Immediately after CT scan of the participant.
  Bone mineral density derived from CT Scan
Bone mineral density Dual-energy x-ray absorptiometry (DXA) | Immediately after DXA scan of the participant.
  Bone mineral density derived from DXA Scan

SECONDARY OUTCOMES:
Correlation between age and bone mineral density | 1 year
  Correlation analysis by means of linear regression and pearson correlation between age (in years) and bone mineral density
Correlation between sex and bone mineral density | 1 year
  Correlation analysis by means of linear regression and pearson correlation between sex (male/female) and bone mineral density
Correlation between height and bone mineral density | 1 year
  Correlation analysis by means of linear regression and pearson correlation between height (in cm) and bone mineral density
Correlation between weight and bone mineral density | 1 year
  Correlation analysis by means of linear regression and pearson correlation between weight and bone mineral density
Correlation between body mass index (BMI) and bone mineral density | 1 year
  Correlation analysis by means of linear regression and pearson correlation between body mass index (BMI, in kg/m^2) and bone mineral density

CONTACTS AND LOCATIONS:
Overall Officials: Hatem Alkadhi, MD, MPH, Principal Investigator — Diagnostic and Interventional Radiology, University Hospital Zurich
Locations (1):
- Diagnostic and Interventional Radiology, University Hospital Zurich, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No